CLINICAL TRIAL: NCT03707808
Title: A Randomized Phase II Clinical Trial on Intratumoral AS01B/ipilimumab Plus Intravenous Nivolumab with or Without Autologous CD1c(BDCA-1)+ / CD141(BDCA-3)+ Myeloid Dendritic Cells.
Brief Title: Intratumoral Injection of Autologous CD1c (BDCA-1)+ MyDC, Avelumab, and Ipilimumab Plus Systemic Nivolumab
Acronym: myDAvIpNi
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-BN-003
Record Dates: First submitted 2018-02-05; First posted 2018-10-16 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-10

CONDITIONS: Solid Tumor; Metastases to Soft Tissue
Keywords: solid tumors
MeSH Terms: interventions — avelumab; Nivolumab

STUDY DESIGN:
Intervention Model Description: There are 2 arms that are given treatment in parallel. But pts from the second arm without the myDC are able to crossover to the first arm with the myDC's. But not the other way around.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate treatment (Experimental): IT injection of MyDC, ipilimumab and AS01b + IV nivolumab
  Interventions: Drug: intratumoral injection of autologous CD1c (BDCA-1)+ myDC; Drug: Intratumoral injection of ipilimumab and AS01b; Drug: IV nivolumab
- Delayed treatment (Active Comparator): IT injection of ipilimumab and AS01b + IV nivolumab
  Interventions: Drug: Intratumoral injection of ipilimumab and AS01b; Drug: IV nivolumab

INTERVENTIONS:
Drug: intratumoral injection of autologous CD1c (BDCA-1)+ myDC — intratumoral injections plus intravenous administration
  Other Names: intratumoral injection of ipilimumab and avelumab; intravenous nivolumab
  Arms: Immediate treatment
Drug: Intratumoral injection of ipilimumab and AS01b — Intratumoral injection of ipilimumab and AS01b
Drug: IV nivolumab — Nivolumab administered intravenously

SUMMARY:
This phase II trial aims at investigating the role and effect of autologous CD1c (BDCA-1)+ myeloid dendritic cells in combination with intratumoral injection of the CTLA-4 blocking monoclonal antibody (mAb) ipilimumab and the immunoligand AS01B compared to a combinatorial immunotherapy regimen using intratumoral injection of the CTLA-4 blocking monoclonal antibody (mAb) ipilimumab and the immunoligand AS01B. Concomitantly, nivolumab (a PD-1 blocking mAb) will be administered intravenously in both arms.

DETAILED DESCRIPTION:
This phase II trial aims at investigating the role and effect of autologous CD1c (BDCA-1)+ myeloid dendritic cells in combination with intratumoral injection of the CTLA-4 blocking monoclonal antibody (mAb) ipilimumab and the immunoligand AS01B compared to a combinatorial immunotherapy regimen using intratumoral injection of the CTLA-4 blocking monoclonal antibody (mAb) ipilimumab and the immunoligand AS01B. Concomitantly, nivolumab (a PD-1 blocking mAb) will be administered intravenously in both arms.

CD1c (BDCA-1)+ myeloid dendritic (myDC) cells will be obtained by immunomagnetic isolation from PBMC obtained by leukapheresis. The CD1c (BDCA-1)+ myDC will not be substantially manipulated prior to autologous intratumoral injection, immediately following the isolation and concentration (isolation and administration will be performed in the same procedure). The investigators consider that the isolation represents a non-substantial manipulation of this somatic cell therapy product. The intended use of CD1c (BDCA-1)+ myDC in this clinical protocol is to enrich their presence within the injected metastasis where they should execute their physiological role of coordinating the anti-tumor immune response. Based on recent preclinical data, absence of myeloid dendritic cells in the tumor microenvironment is an important immune escape mechanism of malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent prior to initiation of any study-specific activities/procedures.
* Male or female age ≥ 18 years at the time of informed consent
* Histologically confirmed advanced solid tumor that cannot be completely surgically resected
* Failing all standard curative and live prolonging therapy.
* Presence of skin- or lymphnode metastatic disease amenable to intratumoral injection by manual palpation, US or CT-guidance. At least one metastatic lesion should be amenable to a safe post-injection biopsy (by core needle biopsy, partial- or complete surgical resection).
* ECOG performance status of 0 or 1
* Candidate for intralesional therapy defined as either one of the following:
* At least 1 injectable skin or lymph node metastatic lesion with a longest diameter of ≥ 10 mm
* Multiple injectable tumor lesions that in aggregate have a longest diameter of ≥ 10 mm injectable disease
* Adequate organ function determined within 14 days prior to enrollment, defined as follows:
* Hematological: absolute neutrophil count ≥ 1500/mm3 (1.5x109/L), platelet count: ≥ 100.000/mm3 (7.5x109/L), hemoglobin: ≥ 9 g/dL (without need for hematopoietic growth factor or transfusion support)
* Renal: serum creatinine: 1.5 x upper limit of normal (ULN), OR 24-hour creatinine clearance ≥ 60 mL/min for subject with creatinine levels > 1.5 x ULN. (Note: Creatinine clearance need not be determined if the baseline serum creatinine is within normal limits. Creatinine clearance should be calculated per institutional standard).
* Hepatic: serum bilirubin: 1.5 x ULN OR direct bilirubin ≤ ULN for a subject with total bilirubin level > 1.5 x ULN, aspartate aminotransferase (AST): 2.5 x ULN OR ≤ 5 x ULN for subject with liver metastases, alanine aminotransferase (ALT): 2.5 x ULN OR ≤ 5 x ULN for subject with liver metastases
* Coagulation: international normalization ratio (INR) or prothrombin time (PT): 1.5 x ULN unless the subject is receiving anticoagulant therapy as long as PT and partial thromboplastin time (PTT)/ activated PTT (aPTT) is within therapeutic range of intended use of anticoagulants, PTT or aPTT: 1.5 x ULN unless the subject is receiving anticoagulant therapy as long as PT and PTT/aPTT is within therapeutic range of intended use of anticoagulants
* Female subject of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to enrollment. If urine pregnancy test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Availability of a tumor sample (archival sample obtained within 3 months prior to study participation or newly obtained biopsy). Subject must submit the tumor sample during screening. Subjects with a non-evaluable archival sample may obtain a new biopsy and subjects with a non-evaluable newly obtained biopsy may undergo re-biopsy at the discretion of the investigator.
* Adequate vascular access to undergo a leucapheresis.

Exclusion Criteria:

* Known active central nervous system (CNS) metastases. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids >8 mg/day of methylprednisone or equivalent. The exception does not include carcinomatosus meningitis which is excluded regardless of clinical stability.
* History or evidence of active autoimmune disease that requires systemic treatment (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* History or evidence of immunodeficiency states (eg, hereditary immune deficiency, organ transplant, or leukemia)
* History of other malignancy within the past 5 years with the following exceptions: malignancy treated with curative intent and with no known active disease present and has not received chemotherapy for > 5 years before enrollment and felt to be at low risk for recurrence by the treating physician, adequately treated non-melanoma skin cancer without evidence of disease at the time of enrollment, adequately treated cervical carcinoma in situ without evidence of disease at the time of enrollment, adequately treated breast ductal carcinoma in situ without evidence of disease at the time of enrollment , prostatic intraepithelial neoplasia without evidence of prostate cancer at the time of enrollment, adequately treated superficial or in-situ carcinoma of the bladder without evidence of disease at the time of enrollment
* Prior treatment of other tumor vaccine
* Prior chemotherapy, radiotherapy, biological cancer therapy, targeted therapy, or major surgery within 28 days prior to enrollment or has not recovered to CTCAE grade 1 or better from adverse event due to cancer therapy administered more than 28 days prior to enrollment.
* Currently receiving treatment in another investigational device or drug study, or less than 28 days since ending treatment on another investigational device or drug study
* Expected to require other cancer therapy while on study with the exception of local radiation treatment to the site of bone and other metastasis for palliative pain management
* Other investigational procedures while participating in this study are excluded.
* History or evidence of symptomatic autoimmune pneumonitis, glomerulonephritis, vasculitis, or other symptomatic autoimmune disease, or active autoimmune disease or syndrome that has required systemic treatment in the past 2 years (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs) except vitiligo or resolved childhood asthma/atopy. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Evidence of clinically significant immunosuppression such as the following: diagnosis of immunodeficiency, concurrent opportunistic infection, receiving systemic immunosuppressive therapy (> 2 weeks) or within 7 days prior to the first dose of study treatment, including oral steroid doses > 10 mg/day of prednisone or equivalent except for management of adverse events and central nervous system (CNS) metastases during the course of the study. Subjects that require intermittent use of bronchodilators or local steroid injection will not be excluded from the study.
* Known human immunodeficiency virus (HIV) disease
* Known acute or chronic hepatitis B or hepatitis C infection
* Female subject is pregnant or breast-feeding, or planning to become pregnant during study treatment and through 3 months after the last dose of study treatment
* Female subject of childbearing potential who is unwilling to use acceptable method(s) of effective contraception during study treatment and through 3 months after the last dose of study treatment. Note: Women not of childbearing potential are defined as: postmenopausal (defined as at least 12 months with no menses without an alternative medical cause; in women < 45 years of age a high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. In the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.) OR have had a hysterectomy and/or bilateral oophorectomy, bilateral salpingectomy or bilateral tubal ligation/occlusion, at least 6 weeks prior to screening; OR has a congenital or acquired condition that prevents childbearing. Note: Acceptable methods of effective contraception are defined in the informed consent form.
* Male subject unwilling to use acceptable method of effective contraception during trial participation and through 3 months after the last dose of study treatment. For this trial, male subjects will be considered to be of non-reproductive potential if they have azoospermia (whether due to having had a vasectomy or due to an underlying medical condition). Note: Acceptable methods of effective contraception are defined in the informed consent form.
* Subject has known sensitivity to any of the products or components to be administered during dosing
* Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the subject and investigator's knowledge
* History or evidence of psychiatric, substance abuse, or any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion
* Is or has an immediate family member (eg, spouse, parent/legal guardian, sibling, or child) who is investigational site or sponsor staff directly involved in the this trial, unless prospective institutional review board (IRB)/independent ethics committee (IEC) approval (by chair or designee) is given allowing exception to this criterion for a specific subject
* Sexually active subject who is unwilling to use a barrier method to avoid potential viral transmission during sexual contact during and within 3 months after study treatment.
* Prior allogeneic hematopoietic stem cell transplantation within the last 5 years. (Subjects who have had a transplant > 5 years ago are eligible as long as there are no symptoms of Graft versus Host Disease.)
* Known history of active Bacillus tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2018-01-29 (Actual); Primary Completion 2025-12-24 (Estimated); Study Completion 2025-12-24 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Treatment-related Adverse Events graded according to CTCAE of intratumoral injection of autologous CD1c (BDCA-1)+ myDC plus avelumab and ipilimumab in combination with iv nivolumab | 1 year
  Participants with treatment-related adverse events will be assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
To assess the therapeutic efficacy and toxicity of the AS01B adjuvants in combination with systemic PD-1 blockade and intratumoral CTLA-4 inhibition plus intratumoral administration of CD1c (BDCA-1)+ / CD141 (BDCA-3)+ myDC co-product in patients | 1 year
  1-year progression free survival (PFS) rate following randomization.
Feasibility of treatment strategy | 1 year
  Percentage of study patients that can receive the planned CD1c (BDCA-1)+ / CD141(BDCA-3)+ myDC intratumoral injection.

SECONDARY OUTCOMES:
Objective response rate (ORR) of intratumoral injected CD1c (BDCA-1)+ myDC, avelumab, and ipilimumab plus iv nivolumab | 1 year
  Objective response rate (ORR, defined as the percentage of subjects with a confirmed complete response (CR), or partial response at any time per Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1
Treatment disposition | 1 year
  Number/volume of administered CD1c (BDCA-1)+ / CD141 (BDCA-3)+ myDC Administered dose of AS01, ipilimumab, and nivolumab
Anti-tumor activity | 1 year
  Tumor response (ORR) according to RECISTv1.1 and iRECIST Tumor response and duration of response of CD1c (BDCA-1)+
  / CD141 (BDCA-3)+ myDC, AS01, and ipilimumab injected and non-injected metastases (reported descriptively)
Duration of response (DOR) | 1 year
  Duration of response of CD1c (BDCA-1)+ / CD141 (BDCA-3)+ myDC, AS01B and ipilimumab in injected and non-injected metastases (reported descriptively)
Progression-free survival (PFS) | 1 year
  Time from first study treatment administration to progression of disease according to RECISTv1.1 and iRECIST (and possibly itRECIST)
Overall survival | 1 year
  Time from first study treatment administration to death

OTHER OUTCOMES:
Effect on cellular- and molecular characteristics of the tumor microenvironment during/following study treatment | 1 year
  Immunohistochemical analysis (CD3, CD8, CD4, PD-L1), multiplexed immunofluorescent imaging, and RNA-expression profiling (NanoString PanCancer IO 360 gene expression panel) of repetitive on-treatment tissue biopsies/FNA of injected metastases T-cell receptor repertoire in metastases assessed by ImmunoSEQ analysis
Effect of study treatment on blood lymphocytes | 1 year
  Peripheral blood differential white blood cell counts Immunocytochemical differential cell counts (incl. CD3+, CD4+ and CD8+ lymphocytes) T-cell receptor repertoire assessed by ImmunoSEQ analysis Flow cytometric analysis of effector/naïve/memory T cells

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tijtgat J, Geeraerts X, Boisson A, Stevens L, Vounckx M, Dirven I, Schwarze JK, Raeymaeckers S, Forsyth R, Van Riet I, Tuyaerts S, Willard-Gallo K, Neyns B. Intratumoral administration of the immunologic adjuvant AS01B in combination with autologous CD1c (BDCA-1)+/CD141 (BDCA-3)+ myeloid dendritic cells plus ipilimumab and intravenous nivolumab in patients with refractory advanced melanoma. J Immunother Cancer. 2024 Jan 11;12(1):e008148. doi: 10.1136/jitc-2023-008148. PMID 38212127